CLINICAL TRIAL: NCT00982774
Title: Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of the LEISH-F2 + MPL-SE Vaccine in Combination With SSG in the Treatment of Patients With PKDL
Brief Title: Safety and Immunogenicity of the LEISH-F2 + MPL-SE Vaccine With SSG for Patients With PKDL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Responsible Party: Professor Eltahir Khalil/PI and Franco Piazza/IDRI Study Director, Institute of Endemic Diseases and Infectious Disease Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IDRI-LVPTC-107
Record Dates: First submitted 2009-09-21; First posted 2009-09-23 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Post Kala Azar Dermal Leishmaniasis
Keywords: PKDL

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: LEISH-F2 + MPL-SE vaccine — LEISH-F2 protein (10 ug) + MPL-SE (25ug) Three injections, 14 days apart

SUMMARY:
A phase 1, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and immunogenicity of three injections of 10 µg LEISH-F2 + 25 µg MPL-SE given at 14-day intervals as an adjunct to standard chemotherapy with sodium stibogluconate (20 mg/kg/day for 40 days) in patients with PKDL.

ELIGIBILITY:
Inclusion Criteria:

* Males and females = 7 years and < 40 years of age.
* Must have a skin rash of > 6 months duration compatible with a diagnosis of PKDL following a history of successful treatment of VL, and histopathology consistent with PKDL (Section 6.1).
* Female patients of child bearing age must have a negative serum pregnancy test at screening, a negative urine pregnancy test within 24 hours before study injection, must not be breast-feeding, and are required to use adequate contraception through Day 59 of the study. These precautions are necessary due to unknown effects that LEISH-F2 + MPL-SE might have in a fetus or newborn infant.
* The following laboratory blood tests must have values within the normal ranges at screening (Appendix 3): sodium, potassium, urea, total bilirubin, glucose, creatinine, hemoglobin and platelet count. ALT, AST, alkaline phosphatase, and total WBC count values (commonly elevated in PKDL patients) must be below grade 2 at screening (Appendix 3).
* The following serology tests must be negative at screening: HIV 1/2 (in patients >14 years of age), hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody. All patients (or their parents) will receive HIV-related counseling prior to testing. Patients with positive HIV test results will receive counseling at the University and will be referred to the national AIDS control program for treatment if appropriate.
* Normal ECG.
* Potential study patients (or their guardians) must give written informed consent, be willing to be admitted to hospital for a minimum of 40 days and up to 60 days, able to attend all required follow-up visits, have a permanent address, and be reachable by study site personnel.

Exclusion Criteria:

* Presence of other skin conditions.
* Anti-leishmanial treatment within the past 30 days.
* History of previous exposure to Leishmania vaccines.
* Known use of injected or oral corticosteroids within 6 weeks prior to the first administration of study injection.
* Participation in another experimental protocol or receipt of any investigational products within 30 days prior to the first administration of study injection.
* History of autoimmune disease or other causes of immunosuppressive states.
* History or evidence of any acute or chronic illness that, in the opinion of the Principal Investigator, may interfere with the evaluation of the safety or the immunogenicity of the vaccine. (Patients presenting with concomitant illness will be referred for standard clinical care).
* History of use of any medication that, in the opinion of the Principal Investigator, may interfere with the evaluation of the safety or the immunogenicity of the vaccine.
* History of significant psychiatric illness.
* Known to be a current drug or alcohol abuser.
* Patients with a history of previous anaphylaxis, severe allergic reaction to vaccines or unknown allergens, or allergic reaction to eggs.
* Patients who are unlikely to cooperate with the requirements of the study protocol.
* Known allergy or contraindication to SSG.
* Regardless of eligibility, standard clinical care will be provided (at no cost to the patient) to all PKDL patients screened for participation in the study.

Ages: 7 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of the vaccine given as 3 sc injections every 14 days in combination with standard SSG therapy in patients with persistent PKDL. | one year

SECONDARY OUTCOMES:
Assess the effect of the vaccine on the clinical course of PKDL. | one year
To evaluate the immunogenicity of the vaccine by evaluating antibody and T-cell responses to the LEISH-F2 protein and Soluble Leishmania Antigen (SLA). | one year

CONTACTS AND LOCATIONS:
Overall Officials: Eltahir AG Khalil, MBBS, Principal Investigator — IEND; Franco Piazza, MD, MPH, Study Director — Access to Advanced Health Institute (AAHI)
Locations (1):
- IEND, Khartoum, Sudan